CLINICAL TRIAL: NCT02228941
Title: NFIL3-induced Pathological Enhancement of IgE Class Switch Recombination in Hyper-IgE Syndrome
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Shanghai Children's Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 81273314
Record Dates: First submitted 2014-08-18; First posted 2014-08-29 (Estimated); Last update posted 2014-08-29 (Estimated); Status verified 2014-08

CONDITIONS: Job Syndrome
MeSH Terms: conditions — Job Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months

GROUPS / COHORTS (1):
- gene mutation

SUMMARY:
Hyper IgE syndrome (HIES) is a rare and complex primary immunodeficiency that affects multiple systems. It is characterized by elevated Immunoglobulin E(IgE), recurrent skin and pulmonary infections and eczematoid dermatitis.Somatic manifestations include scoliosis, joint hyperextensibility, impaired shedding of deciduous teeth and facial dysmorphism.

The reason of extremely high level of serum IgE in the patients with HIES is unknown. Signal transducers and activators of transcription 3(STAT3) gene mutations can cause the STAT3/Janus kinase(STAT3/JAK) signal transduction pathway disorder, then can affect the B cell development.

It is reported that levels of extracellular signal cytokine and the prolonged half-life of IgE are not the causes of dramatically increased IgE levels in STAT3-HIES patients. According to our preliminary work, we found that the slight increase of IgE-secreting plasma cells could not explain the tremendously increased IgE level and that the key class switch recombination enzyme (AID) was up-regulated in STAT3-HIES patients. Intriguingly, we found that deregulation of immunoglobulin class switch recombination (CSR) in IgE secreting plasma cells in STAT3-HIES patients might play a key role in dramatically increased IgE levels.

Nuclear factor IL-3 regulated (NFIL3) is a newly discovered transcriptional factor. During STAT3-HIES IgE-secreting plasma cells differentiating, NFIL3 was significantly upregulated. The CSR of IgE was down-regulated in STAT3-deficiency mice as well as NFIL3-deficiency mice, however Interleukin-4（IL-4）, a STAT3-independent cytokine, promotes NFIL3 expression by Signal transducers and activators of transcription 6(STAT6) dependent manner. Thus, we hypothesize that NFIL3 may play a key role in dramatically increased IgE levels in STAT3-HIES patients.

In-depth insight of the pathogenic role of NFIL3 within human STAT3-HIES has great significance in clarifying the pathogenesis of HIES and exploiting effective targeting interventions to improve clinical outcomes. Also, it can provide valuable clues for the clinical treatment of IgE-related diseases, such as parasite infection and malignant diseases.

ELIGIBILITY:
Inclusion Criteria:

* Group 1 AD-HIES patients A.Patients with extremely high serum IgE levels, IgE>2000IU/ml; B.Patients diagnosis referred to the NIH, and NIH score>15; C.Patients must be confirmed with clinical manifestations of AD-HIES, namely:skin abscesses,pneumonias,distinctive facial appearance,dental abnormalities,minimal trauma fractures D.Patients must be confirmed with STAT3 gene mutations;
* Group 2 AR-HIES patients A.Patients with extremely high serum IgE levels, IgE>2000IU/ml; B.Patients diagnosis referred to the NIH, and NIH score>15; C.Patients must be confirmed with clinical manifestations of AR-HIES, namely:pneumonias,eczema,Skin abscesses,mucocutaneous viral infections,malignancy D.Patients must be confirmed with Dedicator of cytokinesis protein 8（DOCK8） or Tyrosine Kinase 2(Tyk2) gene mutations;
* Group 3 Healthy Control A.Healthy control aged 1-25 year at time of enrollment.

Exclusion Criteria for all groups:

* Any subjects with serious conditions requiring treatment or hospitalization;
* Any subjects with pregnancy;
* Any subjects who have a history of bone marrow transplant,or have received treatment with chemotherapy or radiation;

Ages: 1 Month to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: We divided the patients with HIES into two groups, namely Autosomal-dominant Hyper-IgE Syndrome(AD-HIES) group and Autosomal-recessive Hyper-IgE Syndrome(AR-HIES) group. According to the different group, we need to do a variety of detection index, for example, gene mutations, B-lymphocyte subsets, protein expression et al.In addition, healthy control group is needed in the experiment.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2014-09; Primary Completion 2014-09 (Estimated)

PRIMARY OUTCOMES:
Times of Pneumonia | 1 year
Times of Skin abscess | 1 year